CLINICAL TRIAL: NCT05883787
Title: Development of a Technical Solution to Digitalize the Analysis of Failure and Effects.
Acronym: e-AMFE
Status: Withdrawn | Type: Observational
Why Stopped: Not enough budget to carry it out.
Sponsor: José Joaquín Mira Solves (Other)
Responsible Party: Sponsor-Investigator, José Joaquín Mira Solves, Professor, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Organization: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Other Study IDs: UGP-22-379
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Notification, Spousal

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Exploration of a database — extraction of data

SUMMARY:
This is a preliminar study to extract information from the data base of health inquiries from the Valencian community and to charge them in the analysis of modules and effects.

ELIGIBILITY:
Inclusion Criteria:

* To be a notification of a health inquiry

Exclusion Criteria:

* None

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients in the Valencian community in Spain
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
FMEA | 1 year
  Failure Mode and Effect Analysis

CONTACTS AND LOCATIONS:
Locations (1):
- FISABIO, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided